CLINICAL TRIAL: NCT05984290
Title: Study to Evaluate Safety and Effectiveness of the Boston Orthokeratology (Oprifocon A) Shaping Lens in the Arise Orthokeratology Lens Design With Non-spherical Posterior Peripheral Curves
Brief Title: Study of Safety and Effectiveness of the Boston Orthokeratology Shaping Lens in the Arise Orthokeratology Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 918
Record Dates: First submitted 2023-08-02; First posted 2023-08-09 (Actual); Results first posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Safety and effectiveness of the Arise Orthokeratology Lens (Experimental): Treatment effect of overnight orthokeratology over a 3-month period
  Interventions: Device: orthokeratology lens

INTERVENTIONS:
Device: orthokeratology lens — Each subject will wear the study lenses in both eyes overnight for approximately 3 months.

SUMMARY:
The objective of this orthokeratology study is to evaluate the safety and effectiveness of the Arise Orthokeratology Lens with non-spherical posterior peripheral curves

DETAILED DESCRIPTION:
The Bausch + Lomb Vision Shaping Treatment VST is based on a reverse geometry orthokeratology design that includes a base curve/treatment curve, a reverse curve, alignment curves and peripheral curves. The base curve is used to only flatten the cornea and is not considered a fitting curve. The parameters of the Arise Orthokeratology Lens are controlled to be within the bounds determined by the spherical posterior curves of other lens designs prescribed for the Bausch + Lomb Vision Shaping Treatment. The term peripheral curves excludes the base curve and includes the zones defined as the reverse curve, alignment curves and peripheral curves. Peripheral curves are designed to help control centration of the lens. When there are elevation differences between the flat and steep meridians on the cornea (e.g., corneal toricity), spherical peripheral curves, including the reverse curve, alignment curves and peripheral curves, may not align completely to the cornea and can result in a lens with sub-optimal centration. Aspheric curves and toric (e.g., dual axis) peripheral curves on reverse geometry lenses for overnight orthokeratology have been available in the US market for more than 10 years for fitting lenses. The intent of the Arise Orthokeratology Lens is to provide a stable and centered lens that helps ensure the treatment zone of the lens is well positioned in relation to the pupil and is shaping the central portion of the cornea for optimal results.

ELIGIBILITY:
Inclusion Criteria:

1. Be 12 years or older on the date the Informed Consent Form (ICF) is signed and, as subject or parent or legal guardian of a minor subject, have capacity to read, understand and provide written voluntary informed consent on the IRB-approved ICF and provide authorization as appropriate for local privacy regulations.
2. Be orthokeratology lens naïve.
3. Spherical refractive error between plano and -5.00D.
4. Astigmatism no greater than 1.50D.
5. Corneal topography sagittal height differential of ≥ 30 microns between the two main meridians (flat and steep) at an 8mm chord.
6. Has keratometric readings from 39.00 to 48.00D.
7. Has a clear and undistorted Mire Reflex.
8. Be willing and able to comply with all treatment and follow-up study visits and procedures.
9. Must be willing to refrain from wearing habitual soft contact lenses during the study period.
10. Subjects must be correctable through spherocylindrical refraction to 42 letters (0.1 logMAR) or better (distance, high contrast) in each eye.

Exclusion Criteria:

1. Subject is considered by the Investigator, to not be a suitable candidate for participation or it is not in the best interest of the subject to participate in the study.
2. Subjects who have worn rigid gas permeable (RGP) contact lenses within the last 30 days or who have worn polymethylmethacrylate (PMMA) lenses within the last three months.
3. Prior eyelid, strabismus, intraocular, or refractive surgery.
4. Keratoconus or an irregular cornea.
5. Subjects with any systemic disease currently affecting ocular health or in the Investigator's opinion may have an effect on ocular health during the course of the study.
6. Subjects using any systemic or topical medications that will, in the Investigator's opinion, affect ocular physiology or lens performance.
7. A known allergy to fluorescein, benoxinate, or proparacaine.
8. A history of corneal hypoesthesia (reduced corneal sensitivity), corneal ulcer, corneal infiltrates, ocular viral or fungal infections or recurrent ocular infections.
9. Subjects with an active ocular disease or who are using any ocular medication.
10. Subjects with any Grade 2 or greater finding during the slit lamp examination. Subjects with corneal infiltrates, of ANY GRADE, are NOT eligible. Refer to Appendix B: Methods of Clinical Evaluation.
11. Subjects with any "Present" finding during the slit lamp examination that, in the Investigator's judgement, interferes with contact lens wear. Refer to Appendix B: Methods of Clinical evaluation.
12. Subjects with any scar or neovascularization within the central 6mm of the cornea. Subjects with minor peripheral corneal scarring (that does not extend into the central area), that in the Investigator's judgement, does not interfere with contact lens wear, are eligible for this study.
13. Subjects participating in any drug or device clinical investigation within 2 weeks prior to entry into this study (Screening Visit) and/or planning to do so during the period of study participation.
14. Subjects who are amblyopic.
15. Immediate family or close relative is a member of the office staff, including the Investigator(s).
16. Females of childbearing potential (those who are not surgically sterilized or postmenopausal) if they meet any one of the following:

    * They are currently pregnant
    * They plan to become pregnant during the study
    * They are breastfeeding

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Levenson Eye Associates, Jacksonville, Florida
  - Birmingham Vision Care P.C., Bloomfield, Michigan
  - Cornea and Contact Lens Institute of Minnesota, Edina, Minnesota
  - The Koetting Associates, St Louis, Missouri
  - Optometric Physicians of Middle Tennessee, Nashville, Tennessee
  - Speciality Eyecare Group, Kirkland, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Groups:
- Safety and Effectiveness of the Arise Orthokeratology Lens: Treatment effect of overnight orthokeratology over a 3-month period orthokeratology lens: Each subject will wear the study lenses in both eyes overnight for approximately 3 months.
Period: Dispensing
Arm/Group | Safety and Effectiveness of the Arise Orthokeratology Lens
Started | 90; 180 Eyes
Completed | 76; 152 Eyes
Not Completed | 14; 28 Eyes
Period: Study Treatment
Arm/Group | Safety and Effectiveness of the Arise Orthokeratology Lens
Started | 76; 152 Eyes
Completed | 46; 92 Eyes
Not Completed | 30; 60 Eyes

BASELINE CHARACTERISTICS:
Arm/Group | Safety and Effectiveness of the Arise Orthokeratology Lens
Number analyzed (Participants) | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (10.72)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 48
  Male | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic and Not Latino | 67
  White | 51
  Black or African American | 10
  Asian | 11
  Multiple | 2
  Unknown or not reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 76

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Serious Adverse Events at the Subject Level
Time Frame: Assessed from dispensing through 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Safety and Effectiveness of the Arise Orthokeratology Lens
Number analyzed (Participants) | 76
Participants | 0

2. Primary Outcome: Percentage of Subjects Who Achieve Monocular Uncorrected Distance Visual Acuity (UDVA) of 20/40 or Better in Both Eyes
Description: Using the high contrast distance UDVA collected at the 3-Month Follow-up Visit, subjects with non-missing Snellen VA of 20/40 or less in both eyes will be classified as "20/40 or Better". Subjects with at least one missing value at the 3-Month Follow-up Visit will not be classified and their classification value will be assigned as a missing value. The denominator for percentages will be the number of non-missing values
Time Frame: Assessed at 3 month follow up visit
Measure: Count of Participants; unit: Participants
Arm/Group | Safety and Effectiveness of the Arise Orthokeratology Lens
Number analyzed (Participants) | 45
Participants | 42

3. Primary Outcome: The Rate of Serious Adverse Events at the Eye Level
Time Frame: Assessed from dispensing through 3 months
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Safety and Effectiveness of the Arise Orthokeratology Lens
Number analyzed (Participants) | 76
Number analyzed (Eyes) | 152
Eyes | 0

ADVERSE EVENTS:
Time Frame: AE data collected over all scheduled follow-up visits approximately 3 months after study lens dispensed
Arm/Group | Safety and Effectiveness of the Arise Orthokeratology Lens
All-Cause Mortality (participants affected / at risk) | 0/76
Serious Adverse Events (participants affected / at risk) | 0/76
Other Adverse Events (participants affected / at risk) | 6/76
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Safety and Effectiveness of the Arise Orthokeratology Lens (N=76)
Corneal abrasion (Injury, poisoning and procedural complications) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT05984290/Prot_SAP_000.pdf